CLINICAL TRIAL: NCT01098487
Title: A Longitudinal 2-year Bone Marrow Study of Eltrombopag Olamine (SB-497115-GR) in Previously Treated Adults, With Chronic Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Brief Title: A Longitudinal 2-year Bone Marrow Study of Eltrombopag in Previously Treated Adults, With Chronic Immune (Idiopathic) Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112940
Record Dates: First submitted 2010-03-25; First posted 2010-04-02 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-02

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: Immune (idiopathic) thrombocytopenic purpura (ITP); bone marrow fibers; eltrombopag olamine; thrombopoietin receptor agonist
MeSH Terms: conditions — Purpura; Purpura, Thrombocytopenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental): Oral eltrombopag once daily, starting dose 50 mg (or 25 mg for subjects of East Asian ancestry).
  Interventions: Drug: Eltrombopag olamine

INTERVENTIONS:
Drug: Eltrombopag olamine — Thrombopoietin receptor agonist

SUMMARY:
A open-label, multi-center 2-year safety study to ascertain the baseline levels of bone marrow fibers in previously treated adults with chronic immune (idiopathic) thrombocytopenic purpura (ITP) and to evaluate the long-term effect of eltrombopag on bone marrow fibers. The study will also describe the long-term safety and tolerability of oral eltrombopag treatment in subjects with chronic ITP.

DETAILED DESCRIPTION:
This is a phase IV, open-label safety study, designed to determine baseline levels of bone marrow fibers in previously treated adults with chronic immune (idiopathic) thrombocytopenic purpura (ITP)and to evaluate the long-term effect of eltrombopag on bone marrow reticulin and/or collagen fibers.

The duration of the screening period is up to 8 weeks. Eltrombopag will be administered for at least 2-years followed by a 4-week follow-up period. Bone marrow biopsies will be performed at screening, after 1-year and 2-years of eltrombopag treatment, and at early withdrawal of treatment. The screening bone marrow biopsy should be performed within 8 weeks of planned start of study medication and the bone marrow biopsy block must be available for central laboratory processing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed and dated a written informed consent and be able to understand and comply with protocol requirements and instructions.
* Adults (≥18 years) diagnosed with chronic ITP according to the American Society for Hematology/British Committee for Standards in Hematology (ASH/BCSH) guidelines [George, 1996; BCSH, 2003; Provan, 2009]. In addition, a peripheral blood smear should support the diagnosis of ITP with no evidence of other disease causative of thrombocytopenia (e.g., pseudo thrombocytopenia, myelofibrosis). The physical examination should not suggest any disease, which may cause thrombocytopenia other than ITP.
* Subjects must be physically eligible for serial bone marrow biopsies and must have a bone marrow biopsy performed during screening, and be willing to remain on the study for at least 2 years with annual bone marrow biopsies.
* Subjects, who previously received eltrombopag or romiplostim, must have completed treatment with these therapies at least 6 months prior to the screening bone marrow biopsy.
* Subjects must have the following clinical chemistry values:
* ALT and AST < 2xULN;
* Bilirubin <1.5xULN (except for Gilbert's Syndrome);
* Subjects are practicing an acceptable method of contraception as specified in the protocol.
* In France, subjects will be eligible for inclusion in this study, only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Subjects with any clinically relevant abnormality, other than ITP, or any other medical condition or circumstance, which in the opinion of the investigator makes the subject unsuitable for participation in the study or suggests another primary diagnosis (e.g., thrombocytopenia is secondary to another disease).
* Subjects with any concurrent malignant disease and/or a recent history of cancer treatment with systemic chemotherapy and/or radiotherapy.

Exception: Subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.

* Subjects with any prior history of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism), AND ≥ two of the following risk factors: hormone replacement therapy, systemic contraception (containing estrogen), smoking, diabetes, hypercholesterolemia, hypertension, cancer, hereditary thrombophilic disorders (e.g., Factor V Leiden, ATIII deficiency, etc), or any family history of arterial or venous thrombosis.
* Subjects with screening bone marrow fibers of either MF Grade 3 using European Consensus scale or Grade 4 using Bauermeister scale.
* Subjects with a QTc >450 msec or > 480 msec for subjects with Bundle Branch Block.
* Female subjects who are nursing or pregnant (positive serum or urine β-human chorionic gonadotrophin (β-hCG) pregnancy test) at screening.
* Subjects treated with an investigational drug (other than a thrombopopoetin-receptor (TPO-R) agonist) within 30 days or five half-lives (whichever is longer) preceding the first dose of eltrombopag in the study. (For romiplostim or eltrombopag, see inclusion criterion #4).
* Subjects treated with any TPO-R agonist other than romiplostim or eltrombopag.
* Subjects with recent history of alcohol/drug abuse as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2010-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- GSK Investigational Site, New York, New York, United States
- Czechia (3):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- France (3):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Pessac
- Germany (4):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Shatin, New Territories, Hong Kong
- Hungary (3):
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Szeged
- India (4):
  - GSK Investigational Site, Ludhiana
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Surat
  - GSK Investigational Site, Vellore
- Italy (4):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Padua, Veneto
  - GSK Investigational Site, Vicenza, Veneto
- Pakistan (2):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
- South Korea (2):
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul

REFERENCES:
- [Derived] Wong RS, Bakshi K, Brainsky A. Thrombophilia in patients with chronic immune thrombocytopenia. Scand J Clin Lab Invest. 2015 Jan;75(1):13-7. doi: 10.3109/00365513.2014.962597. Epub 2014 Oct 9. PMID 25296772

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 167 participants were enrolled and received at least one dose of study medication. The 5 enrolled participants from center 082877 were excluded from the analysis due to the following: serious good clinical practice (GCP) findings related to informed consent, source documents and investigator study oversight.
Groups:
- Eltrombopag: Participants received an Open-label treatment of eltrombopag administered as a tablet for up to 2 years (104 weeks), followed by a follow-up period of up to 6 months (only 4 weeks for most participants). The starting dose of eltrombopag was 50 milligrams (mg), once daily (QD). East Asian participants started at a dose of 25 mg QD. The maximum dose allowed was 75 mg daily. Dose modifications were allowed based upon each participant's individual platelet count response.
Period: Overall Study
Arm/Group | Eltrombopag
Started | 162
Completed | 118
Not Completed | 44
Not completed — Adverse Event | 22
Not completed — Lack of Efficacy | 11
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: All Treated Subjects (ATS) Population: all participants who received at least one dose of study medication excluding the 5 participants from Center 082877.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] — All Treated Subjects (ATS) Population: all participants who received at least one dose of study medication excluding the 5 participants from Center 082877.
  Years | 43.1 (16.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 58
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Central/South Asian Heritage | 47
  Asian - East Asian Heritage | 32
  Asian - South East Asian Heritage | 1
  White - White/Caucasian/European Heritage | 81
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bone Marrow (BM) Fibers of MF Grade 0, 1, 2 and 3 on the European Consensus (EC) Scale at Baseline
Description: The evaluation of fibrosis was performed using BM biopsies in which the amount of fibrosis was assessed by the EC Grading Scale. This method distinguishes four degrees of fibrosis (myelofibrosis [MF]-0 to MF-3). MF Grade (G) 0 is scattered linear reticulin with no intersections (cross-overs) corresponding to normal BM; MF Grade 1 is loose network of reticulin with many intersections, especially in perivascular areas; MF Grade 2 is diffuse and dense increase in reticulin with extensive intersections, occasionally with only focal bundles of collagen and/or focal osteosclerosis; MF Grade 3 is diffuse and dense increase in reticulin with extensive intersections with coarse bundles of collagen, often associated with significant osteosclerosis. Baseline is defined as the most recent centrally-reviewed BM biopsy prior to first dose of eltrombopag in the study.
Time Frame: Baseline
Population: All Treated Subjects (ATS) Population: all participants who received at least one dose of study medication excluding the 5 participants from Center 082877. Participants with bone marrow biopsy data available in the relevant time period were included.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 159
Participants
  MF-0 | 150
  MF-1 | 9
  MF-2 | 0
  MF-3 | 0

2. Primary Outcome: Number of Participants With a Positive or Negative Collagen Level at Baseline
Description: The number of participants with a positive or negative collagen level was analyzed. Baseline is defined as the most recent centrally-reviewed BM biopsy prior to first dose of eltrombopag in the study.
Time Frame: Baseline
Population: ATS Population. Participants with bone marrow biopsy data available in the relevant time period were included.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 159
Participants
  Negative | 159
  Positive | 0

3. Primary Outcome: Number of Participants With Indicated Grade Change From Baseline in the EC Grading Scale at 1 Year
Description: The change from baseline to on-treatment assessments of European Consensus (EC) scale was analyzed. On-treatment is defined as during the treatment period (including dose interruptions) and up to 14 days after the end of the treatment period. MF-0 is scattered linear reticulin with no intersections (cross-overs) corresponding to normal BM; MF-1 is loose network of reticulin with many intersections, especially in perivascular areas; MF-2 is diffuse and dense increase in reticulin with extensive intersections, occasionally with only focal bundles of collagen and/or focal osteosclerosis; MF-3 is diffuse and dense increase in reticulin with extensive intersections with coarse bundles of collagen, often associated with significant osteosclerosis. Baseline is defined as the most recent centrally-reviewed BM biopsy prior to first dose of eltrombopag in the study.
Time Frame: Baseline and 1 year
Population: ATS Population. Participants with bone marrow biopsy data available in the relevant time period were included.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 127
Participants
  MF-0 to MF-0 | 82
  MF-0 to MF-1 | 33
  MF-0 to MF-2 | 2
  MF-0 to MF-3 | 2
  MF-1 to MF-0 | 3
  MF-1 to MF-1 | 2
  MF-1 to MF-2 | 1
  MF-1 to MF-3 | 0
  MF-2 to MF-0 | 0
  MF-2 to MF-1 | 0
  MF-2 to MF-2 | 0
  MF-2 to MF-3 | 0
  MF-3 to MF-0 | 0
  MF-3 to MF-1 | 0
  MF-3 to MF-2 | 0
  MF-3 to MF-3 | 0
  Missing to MF-0 | 2
  Missing to MF-1 | 0
  Missing to MF-2 | 0
  Missing to MF-3 | 0

4. Primary Outcome: Number of Participants With Indicated Change From Baseline in the EC Grading Scale at 2 Years
Description: as for outcome 3
Time Frame: Baseline and 2 years
Population: ATS Population. Participants with bone marrow biopsy data available in the relevant time period were included.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 93
Participants
  MF-0 to MF-0 | 79
  MF-0 to MF-1 | 9
  MF-0 to MF-2 | 0
  MF-0 to MF-3 | 0
  MF-1 to MF-0 | 2
  MF-1 to MF-1 | 1
  MF-1 to MF-2 | 0
  MF-1 to MF-3 | 0
  MF-2 to MF-0 | 0
  MF-2 to MF-1 | 0
  MF-2 to MF-2 | 0
  MF-2 to MF-3 | 0
  MF-3 to MF-0 | 0
  MF-3 to MF-1 | 0
  MF-3 to MF-2 | 0
  MF-3 to MF-3 | 0
  Missing to MF-0 | 2
  Missing to MF-1 | 0
  Missing to MF-2 | 0
  Missing to MF-3 | 0

5. Primary Outcome: Number of Participants With a Positive or Negative Collagen Level at 1 Year
Description: The change from Baseline to on-treatment assessments of collagen level was analyzed. On-treatment is defined as during the treatment period (including dose interruptions) and up to 14 days after the end of the treatment period.
Time Frame: 1 year
Population: ATS Population. Participants with bone marrow biopsy data available in the relevant time period were included.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 127
Participants
  Negative to Negative | 120
  Negative to Positive | 5
  Positive to Negative | 0
  Positive to Positive | 0
  Missing to Negative | 2
  Missing to Positive | 0

6. Primary Outcome: Number of Participants With a Positive or Negative Collagen Level at 2 Year
Description: as for outcome 5
Time Frame: 2 years
Population: ATS Population. Participants with bone marrow biopsy data available in the relevant time period were included.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 93
Participants
  Negative to Negative | 90
  Negative to Positive | 1
  Positive to Negative | 0
  Positive to Positive | 0
  Missing to Negative | 2
  Missing to Positive | 0

7. Secondary Outcome: Number of Participants With the Indicated Maximum Toxicity Grade for the Indicated Clinical Chemistry Parameters at Any Time Post-Baseline During the Study
Description: Clinical chemistry parameters were summarized according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0: G0, none; G1, mild; G2, moderate; G3, severe; G4, life-threatening or disabling. Clinical chemistry parameters included: albumin, alkaline phosphatase (ALP), alanine amino transferase (ALT), aspartate amino transferase (AST), total bilirubin, calcium (hypercalcemia), calcium (hypocalcemia), potassium (hyperkalemia), potassium (hypokalemia), sodium (hypernatremia), sodium (hyponatremia), inorganic phosphorus and creatinine. Baseline values were obtained at Day 1. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). The maximum post-Baseline toxicity grade includes any scheduled or unscheduled post-Baseline assessment during.
Time Frame: From Week 1 up to Week 104 and up to 6 months follow-up (4 weeks for most participants) (up to approximately 2.5 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 162
Participants
  Albumin, G0, n=162 | 151
  Albumin, G1, n=162 | 5
  Albumin, G2, n=162 | 6
  Albumin, G3, n=162 | 0
  Albumin, G4, n=162 | 0
  ALP, G0, n=162 | 125
  ALP, G1, n=162 | 35
  ALP, G2, n=162 | 2
  ALP, G3, n=162 | 0
  ALP, G4, n=162 | 0
  ALT, G0, n=162 | 109
  ALT, G1, n=162 | 37
  ALT, G2, n=162 | 8
  ALT, G3, n=162 | 7
  ALT, G4, n=162 | 1
  AST, G0, n=162 | 99
  AST, G1, n=162 | 48
  AST, G2, n=162 | 8
  AST, G3, n=162 | 5
  AST, G4, n=162 | 2
  Total bilirubin, G0, n=162 | 103
  Total bilirubin, G1, n=162 | 40
  Total bilirubin, G2, n=162 | 17
  Total bilirubin, G3, n=162 | 2
  Total bilirubin, G4, n=162 | 0
  Calcium (hypercalcemia), G0, n=162 | 159
  Calcium (hypercalcemia), G1, n=162 | 2
  Calcium (hypercalcemia), G2, n=162 | 1
  Calcium (hypercalcemia), G3, n=162 | 0
  Calcium (hypercalcemia), G4, n=162 | 0
  Calcium (hypocalcemia), G0, n=162 | 92
  Calcium (hypocalcemia), G1, n=162 | 57
  Calcium (hypocalcemia), G2, n=162 | 12
  Calcium (hypocalcemia), G3, n=162 | 0
  Calcium (hypocalcemia), G4, n=162 | 1
  Potassium (hyperkalemia), G0, n=162 | 138
  Potassium (hyperkalemia), G1, n=162 | 14
  Potassium (hyperkalemia), G2, n=162 | 5
  Potassium (hyperkalemia), G3, n=162 | 5
  Potassium (hyperkalemia), G4, n=162 | 0
  Potassium (hypokalemia), G0, n=162 | 123
  Potassium (hypokalemia), G1, n=162 | 35
  Potassium (hypokalemia), G2, n=162 | 0
  Potassium (hypokalemia), G3, n=162 | 4
  Potassium (hypokalemia), G4, n=162 | 0
  Sodium (hypernatremia), G0, n=162 | 138
  Sodium (hypernatremia), G1, n=162 | 20
  Sodium (hypernatremia), G2, n=162 | 2
  Sodium (hypernatremia), G3, n=162 | 2
  Sodium (hypernatremia), G4, n=162 | 0
  Sodium (hyponatremia), G0, n=162 | 137
  Sodium (hyponatremia), G1, n=162 | 21
  Sodium (hyponatremia), G2, n=162 | 0
  Sodium (hyponatremia), G3, n=162 | 3
  Sodium (hyponatremia), G4, n=162 | 1
  Inorganic phosphorus, G0, n=162 | 100
  Inorganic phosphorus, G1, n=162 | 0
  Inorganic phosphorus, G2, n=162 | 52
  Inorganic phosphorus, G3, n=162 | 10
  Inorganic phosphorus, G4, n=162 | 0
  Creatinine, G0, n=162 | 149
  Creatinine, G1, n=162 | 8
  Creatinine, G2, n=162 | 3
  Creatinine, G3, n=162 | 0
  Creatinine, G4, n=162 | 2

8. Secondary Outcome: Number of Participants With the Indicated Maximum Toxicity Grade for the Indicated Hematology Parameters at Any Time Post-Baseline During the Study
Description: Hematology parameters were summarized according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0: G0, none; G1, mild; G2, moderate; G3, severe; G4, life-threatening or disabling. Hematology parameters included: hemoglobin (increased), hemoglobin (anemia), lymphocyte count (increased), lymphocyte count (decreased), total absolute neutrophil count (ANC), platelet count and white blood cell (WBC) count. Baseline values were obtained at Day 1. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). The maximum post-Baseline toxicity grade includes any scheduled or unscheduled post-Baseline assessment during.
Time Frame: From Week 1 up to Week 104 and up to 6 months follow-up (4 weeks for most participants) (up to approximately 2.5 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 162
Participants
  Hemoglobin (increased), G0, n=162 | 143
  Hemoglobin (increased), G1, n=162 | 17
  Hemoglobin (increased), G2, n=162 | 1
  Hemoglobin (increased), G3, n=162 | 1
  Hemoglobin (increased), G4, n=162 | 0
  Hemoglobin (anemia), G0, n=162 | 55
  Hemoglobin (anemia), G1, n=162 | 63
  Hemoglobin (anemia), G2, n=162 | 31
  Hemoglobin (anemia), G3, n=162 | 13
  Hemoglobin (anemia), G4, n=162 | 0
  Lymphocyte count (increased), G0, n=161 | 122
  Lymphocyte count (increased), G1, n=161 | 0
  Lymphocyte count (increased), G2, n=161 | 39
  Lymphocyte count (increased), G3, n=161 | 0
  Lymphocyte count (increased), G4, n=161 | 0
  Lymphocyte count (decreased), G0, n=161 | 86
  Lymphocyte count (decreased), G1, n=161 | 36
  Lymphocyte count (decreased), G2, n=161 | 26
  Lymphocyte count (decreased), G3, n=161 | 13
  Lymphocyte count (decreased), G4, n=161 | 0
  Total ANC, G0, n=161 | 140
  Total ANC, G1, n=161 | 12
  Total ANC, G2, n=161 | 3
  Total ANC, G3, n=161 | 3
  Total ANC, G4, n=161 | 3
  Platelet count, G0, n=162 | 2
  Platelet count, G1, n=162 | 8
  Platelet count, G2, n=162 | 3
  Platelet count, G3, n=162 | 26
  Platelet count, G4, n=162 | 123
  WBC, G0, n=162 | 135
  WBC, G1, n=162 | 21
  WBC, G2, n=162 | 3
  WBC, G3, n=162 | 3
  WBC, G4, n=162 | 0

9. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) Started On-therapy + 1 Day, >1 to 30 Days Post Therapy and >30 Days Post Therapy
Description: On-therapy + 1 day is defined as AEs started between the first dose of eltrombopag and up to the day after the last dose of eltrombopag; >1 to 30 days post therapy is defined as AEs that started more than 1 day and up to 30 days after the last dose of eltrombopag; >30 days post therapy is defined as AEs started that started more than 30 days after the last dose of eltrombopag. An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, or is a congenital anomaly or birth defect. Medical or scientific judgment should be exercised in other situations.
Time Frame: From Week 1 up to Week 104 and up to 6 months follow-up (4 weeks for most participants) (up to approximately 2.5 years)
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 162
Participants
  Any AE, on-therapy + 1 day | 141
  Any SAE, on-therapy + 1 day | 41
  Any AE, >1 to 30 days post therapy | 12
  Any SAE, >1 to 30 days post therapy | 5
  Any AE, >30 days post therapy | 9
  Any SAE, >30 days post therapy | 1

ADVERSE EVENTS:
Time Frame: On-treatment SAEs and non-serious AEs are defined as events occuring from the start of the treatment (Day 1) up to Week 104 and including the follow-up period of up to 6 months (only 4 weeks for most participants) (up to approximately 2.5 years).
Description: SAEs and non-serious AEs were collected in participants of the ATS Population, comprised of all participants who had received at least one dose of study medication.
Arm/Group | Eltrombopag
Serious Adverse Events (participants affected / at risk) | 42/162
Other Adverse Events (participants affected / at risk) | 114/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=162)
Anaemia (Blood and lymphatic system disorders) | 2
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Adrenal insufficiency (Endocrine disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Gingival bleeding (Gastrointestinal disorders) | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Fatigue (General disorders) | 2
Gait disturbance (General disorders) | 1
Local swelling (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cholecystitis infective (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gallbladder empyema (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Sialoadenitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Hepatic enzyme increased (Investigations) | 2
Liver function test abnormal (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral venous thrombosis (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
Transverse sinus thrombosis (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Psychosomatic disease (Psychiatric disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=162)
Anaemia (Blood and lymphatic system disorders) | 11
Iron deficiency anaemia (Blood and lymphatic system disorders) | 9
Vertigo (Ear and labyrinth disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 21
Dyspepsia (Gastrointestinal disorders) | 16
Gingival bleeding (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 15
Asthenia (General disorders) | 9
Fatigue (General disorders) | 15
Influenza like illness (General disorders) | 15
Pain (General disorders) | 9
Pyrexia (General disorders) | 18
Nasopharyngitis (Infections and infestations) | 17
Upper respiratory tract infection (Infections and infestations) | 20
Viral infection (Infections and infestations) | 13
Contusion (Injury, poisoning and procedural complications) | 11
Alanine aminotransferase increased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 12
Decreased appetite (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 22
Back pain (Musculoskeletal and connective tissue disorders) | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 30
Menorrhagia (Reproductive system and breast disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16
Petechiae (Skin and subcutaneous tissue disorders) | 17
Pruritus (Skin and subcutaneous tissue disorders) | 12
Purpura (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 9
Haematoma (Vascular disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.